CLINICAL TRIAL: NCT01487018
Title: Evaluation of the Application of Point-to-Point Computer-Assisted Navigation for Mirroring-Reconstructing of Unilateral Posttraumatic Zygomatic Deformity: A Randomized Controlled Trial
Brief Title: Evaluation of Navigation Assisted Reconstruction of Posttraumatic Zygomatic Deformity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Gong Xi, Department of Oral and Maxillofacial Surgery, Peking University School and Hospital of Stomatology, Peking University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: gongx31480528
Record Dates: First submitted 2011-11-29; First posted 2011-12-07 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Zygomatic Fractures
Keywords: Zygomatic Fractures; Surgery, Computer-Assisted; Facial Asymmetry
MeSH Terms: conditions — Zygomatic Fractures; Facial Asymmetry | interventions — Surgery, Computer-Assisted; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Navigation Surgery (Experimental): To evaluate the feasibility and accuracy of a new method for planning and realizing zygomatic osteotomies in cases of established post-traumatic deformities using computer assisted navigation.
  Interventions: Procedure: Navigation Surgery
- Traditional Surgery (Active Comparator): To compare with the experimental arm.
  Interventions: Procedure: Traditional Surgery

INTERVENTIONS:
Procedure: Navigation Surgery — To evaluate the feasibility and accuracy of a new method for planning and realizing zygomatic osteotomies in cases of established post-traumatic deformities using computer assisted navigation.
  Other Names: Computer-Aided Surgery; Surgical Navigation
  Arms: Navigation Surgery
Procedure: Traditional Surgery — To compare with the experamental group.
  Other Names: Control Group
  Arms: Traditional Surgery

SUMMARY:
Treatment of late deformities following fractures of the orbitozygomaticomaxillary complex can be considered a formidable challenge, even to the skilled surgeon. However, the development of Computer-Assisted Navigation technology Offers new opportunities in the treatment of such deformities. With the help of navigation system,pre- and intraoperatively,the objective of any supporting medical device for reconstruction of the orbitozygomaticomaxillary complex would be visualization of the real and desired positions of the zygoma. In this randomized controlled trial, the investigators would like to evaluate the feasibility and accuracy of a new method for planning and realizing zygomatic osteotomies in cases of established post-traumatic deformities using computer assisted navigation.

DETAILED DESCRIPTION:
Treatment of late deformities following fractures of the orbitozygomaticomaxillary complex can be considered a formidable challenge. Even to the skilled surgeon, over-or underestimation of the displacement is likely to occur, leading to an unsatisfactory result caused by over- or undercorrection.However,The development of Computer-Assisted Navigation technology Offers new opportunities in the treatment of such deformities. With the help of navigation system,pre- and intraoperatively,the objective of any supporting medical device for reconstruction of the orbitozygomaticomaxillary complex would be visualization of the real and desired positions of the zygoma. In this randomized controlled trial, we would like to evaluate the feasibility and accuracy of a new method for planning and realizing zygomatic osteotomies in cases of established post-traumatic deformities using computer assisted navigation.

ELIGIBILITY:
Inclusion Criteria:

1. post-traumatic unilateral deformities of the zygomaticomaxillary complex
2. The interval after the primary injury should be more than 21 days
3. Meet the operation indication
4. Voluntarily join this study with informed consents

Exclusion Criteria:

1. Obviously asymmetric of craniofacial structure
2. Poor compliance of patient
3. Any other condition that do not fit to participate in the study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Zygomatic Symmetry | 1 month
  Measurement the zygomatic symmetry of postoperative CT scan

SECONDARY OUTCOMES:
Accuracy evaluation of CT image | 1 month
  Anatomic contour of pre-operation design affected side was superimposed on postoperative one. Discrepancy between preoperative simulation and postoperative result was calculated.
Facial Symmetry | 3 month
  Facial symmetry on the Visual Analog Scale and three-dimensional camera

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Professor, Principal Investigator — Department of Oral and Maxillofacial Surgery, Peking University School and Hospital of Stomatology
Locations (1):
- Department of Oral and Maxillofacial Surgery, Peking University School and Hospital of Stomatology, Beijing, China